CLINICAL TRIAL: NCT02708290
Title: Mental Imagery Therapy for Autism (MITA) - an Early Intervention Computerized Language Training Program for Children With ASD
Status: Completed | Type: Observational
Sponsor: ImagiRation, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MITA001
Record Dates: First submitted 2016-03-01; First posted 2016-03-15 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Autistic Disorder; Autism; ASD
MeSH Terms: conditions — Autistic Disorder | interventions — Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test arm: The test group included participants who completed more than one thousand exercises and made no more than one error per exercise.
  Interventions: Other: MITA Prefrontal Synthesis exercises - each activity adapts to deliver the exercise that is at the exact level of difficulty appropriate for a child at any given point in time
- Control arm: The control group included the rest of participants. The test group participants were matched to the control group by age, gender, expressive language, receptive language, sociability, cognitive awareness, and health at the 1st evaluation.
  Interventions: Other: MITA Prefrontal Synthesis exercises - each activity adapts to deliver the exercise that is at the exact level of difficulty appropriate for a child at any given point in time

INTERVENTIONS:
Other: MITA Prefrontal Synthesis exercises - each activity adapts to deliver the exercise that is at the exact level of difficulty appropriate for a child at any given point in time — Mental Imagery Therapy for Autism (MITA) is an early-intervention application for children with Autism Spectrum Disorder (ASD). MITA app uses adaptive-learning technologies, with fun, educational exercises that adapt to a child's abilities, resulting in a highly-customized learning experience. The MITA application is available for free in the Apple Store, Google Play, and Amazon App Store.
  MITA verbal activities start with simple vocabulary-building exercises and progress toward exercises aimed at higher forms of language, such as noun-adjective combinations, spatial prepositions, recursion, and syntax. All exercises are deliberately limited to as few nouns as possible since the aim is not to expand a child's one-word vocabulary, but rather to teach him/her to integrate mental objects in novel ways by utilizing prefrontal synthesis (PFS). MITA activities outside of the verbal domain aim to provide the same PFS training visually through implicit instructions.

SUMMARY:
Mental Imagery Therapy for Autism (MITA) is a unique, early-intervention application for children with Autism Spectrum Disorder (ASD). The app includes bright, interactive puzzles designed to help children learn how to mentally integrate multiple features of an object, an ability that has proven to lead to vast improvements in general learning. Success with MITA puzzles could overtime result in significant improvements in a child's overall development, specifically in the realms of language, attention and visual skills.

SCIENCE BEHIND THE PROJECT:

MITA verbal activities start with simple vocabulary-building exercises and progress towards exercises aimed at higher forms of language, such as noun-adjective combinations, spatial prepositions, recursion, and syntax. For example, a child can be instructed to select the {small/large} {red/ blue/green/orange} ball or to put the cup {on/under/behind/in front of} the table. All exercises are deliberately limited to as few nouns as possible since the aim is not to expand a child's one-word vocabulary, but rather to teach him/her to integrate mental objects in novel ways using active imagination.

MITA nonverbal activities aim to provide the same active imagination training visually through implicit instructions. E.g., a child can be presented with two separate images of a train and a window pattern, and a choice of complete trains. The task is to find the correct complete train and place it into the empty square. This exercise requires not only attending to a variety of different features in both the train and its windows, but also combining two separate pieces into a single image (in other words, mentally integrating separate train parts into a single unified gestalt). As levels progress, the exercises increase in difficulty, requiring attention to more and more features and details. Upon attaining the most difficult levels, the child must attend to as many as eight features simultaneously. Previous results from our studies have demonstrated that children who cannot follow the explicit verbal instruction can often follow an equivalent command implicit in the visual set-up of the puzzle.

As a child progresses through MITA's systematic exercises, he or she is developing the ability to simultaneously attend to a greater number of features, reducing the propensity towards tunnel vision, and thus developing an essential component of language. The ability to mentally build an image based on a combination of multiple features is absolutely necessary for understanding syntax, spatial prepositions and verb tenses.

MITA is designed for early childhood and intended for long-term, daily use. It is designed to be engaging and educational, as well as adaptive and responsive to the individual abilities of each child.

ELIGIBILITY:
Inclusion Criteria:

Autism Spectrum Disorder

Exclusion Criteria:

none

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Autism Spectrum Disorder
Sampling Method: Non-Probability Sample
Enrollment: 6454 (Actual)
Dates: Start 2015-09; Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Andrey Vyshedskiy, Ph.D., Principal Investigator — ImagiRation, LLC
Locations (1):
- ImagiRation LLC, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dunn & Vyshedskiy (2015). Mental Imagery Therapy for Autism (MITA)-an early intervention computerized brain training program for children with ASD. Autism Open Access; 5(3)
- [Background] Rimland, B. & Edelson, S. Autism Research Institute. Autism Treat. Eval. Checkl. ATEC (1999)
- [Background] Braverman J, Dunn R, Vyshedskiy A. Development of the Mental Synthesis Evaluation Checklist (MSEC): A Parent-Report Tool for Mental Synthesis Ability Assessment in Children with Language Delay. Children (Basel). 2018 May 20;5(5):62. doi: 10.3390/children5050062. PMID 29783788
- See also: ImagiRation website with links to MITA download — http://imagiration.com/autism/
- See also: A peer-reviewed article describing MITA — http://goo.gl/lyHw95
- See also: MITA download for iPad and iPhone — https://apps.apple.com/us/app/id1020290425
- See also: MITA download for Amazon Kindle Fire — http://www.amazon.com/Mental-Imagery-Therapy-Autism-MITA/dp/B012P1OX36
- See also: MITA download for Android tablet or smartphone — https://play.google.com/store/apps/details?id=com.imagiration.mita
- See also: MITA FAQs — http://imagiration.com/autism/mita-faqs/
- See also: MITA Testimonials — http://imagiration.com/autism/testimonials-for-mita/
- See also: MITA News — http://imagiration.com/autism/mita-news/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: MITA was made available gratis at all app stores from 2015 to 2020. From this pool of potential study participants, we selected participants for the observation clinical study based on the following criteria:
  1. Consistency: at least three ATEC evaluations completed.
  2. The interval between the first and the last evaluation was six months or longer.
  3. Diagnosis: ASD
  4. Age: 2 to 12 years
  This resulted in 6454 participants, from whom we have selected the test and control groups
Groups:
- Test Arm: Completed More Than One Thousand Exercises: The test group (assigned at the end of the three-year study) included participants who demonstrated engagement with the intervention by completing more than one thousand MITA exercises and making no more than one error per exercise.
  MITA imagination exercises - each activity adapts to deliver the exercise that is at the exact level of difficulty appropriate for a child at any given point in time: Mental Imagery Therapy for Autism (MITA) is an early-intervention application for children with Autism Spectrum Disorder (ASD). MITA app uses adaptive-learning technologies, with fun, educational exercises that adapt to a child's abilities, resulting in a highly-customized learning experience. The MITA application is available for free in the Apple Store, Google Play, and Amazon App Store.
- Control Arm: the Rest of Participants: The control group (assigned at the end of the three-year study) included the participants matched by age, gender, expressive language, receptive language, sociability, cognitive awareness, and health score at the 1st evaluation to the test group participants. The participants that were not matched to the test group were not included into the comparison between the groups.
Period: Overall Study
Arm/Group | Test Arm: Completed More Than One Thousand Exercises | Control Arm: the Rest of Participants
Started | 1009 | 1009
Completed | 1009 | 1009
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Arm: The test group included participants who completed more than one thousand MITA exercises and made no more than one error per exercise.
  MITA imagination exercises - each activity adapts to deliver the exercise that is at the exact level of difficulty appropriate for a child at any given point in time: Mental Imagery Therapy for Autism (MITA) is an early-intervention application for children with Autism Spectrum Disorder (ASD). MITA app uses adaptive-learning technologies, with fun, educational exercises that adapt to a child's abilities, resulting in a highly-customized learning experience. The MITA application is available for free in the Apple Store, Google Play, and Amazon App Store.
- Total: Total of all reporting groups
Arm/Group | Test Arm | Control Arm | Total
Number analyzed (Participants) | 1009 | 1009 | 2018
Age, Customized [Count of Participants; unit: Participants] | 1009 | 1009 | 2018
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 252 | 514
  Male | 747 | 757 | 1504
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Language as Measured by Autism Therapy Evaluation Checklist (ATEC) and Mental Synthesis Evaluation Checklist (MSEC).
Description: Parents complete children's evaluations every three-month. These regular assessments evaluate children over 5 orthogonal subscales. In all subscales a lower score indicates lower severity of ASD symptoms and a higher score indicates more severe symptoms of ASD:
  1. Receptive Language (range: 0 to 40 points; based on MSEC evaluation described in Braverman, J. et.al.)
  2. Expressive Language (range 0 to 28 points; based on ATEC evaluation subscale 1 described in Rimland, B. et al.)
  3. Sociability (range: 0 to 40 points; based on ATEC evaluation subscale 2)
  4. Cognitive Awareness (range: 0 to 36 points; based on ATEC evaluation subscale 3)
  5. Health (range: 0 to 75 points; based on ATEC evaluation subscale 4)
Time Frame: up to three years, assessed at 3 months intervals
Population: The framework for evaluation of score changes over time was explained in Mahapatra et al. Autism Dev Disord, 2018. In short, changes in the score were modeled by applying the Linear Model with repeated measures. Least squares means differences generated by the model are reported below. Participants were matched using propensity score analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Test Arm: The test group included participants who completed more than one thousand exercises and made no more than one error per exercise.
  MITA imagination exercises - each activity adapts to deliver the exercise that is at the exact level of difficulty appropriate for a child at any given point in time: Mental Imagery Therapy for Autism (MITA) is an early-intervention application for children with Autism Spectrum Disorder (ASD). MITA app uses adaptive-learning technologies, with fun, educational exercises that adapt to a child's abilities, resulting in a highly-customized learning experience. The MITA application is available for free in the Apple Store, Google Play, and Amazon App Store.
Arm/Group | Test Arm | Control Arm
Number analyzed (Participants) | 1009 | 1009
units on a scale
  Receptive Language improvement over 3 years | 8.49 (0.65) | 4.87 (0.85)
  Expressive Language improvement over three years | 5.03 (0.43) | 3.53 (0.57)
  Sociability improvement over 3 years | 1.88 (0.59) | 0.72 (0.78)
  Cognitive Awareness improvement over 3 years | 2.43 (0.52) | 2.19 (0.68)
  Health improvement over 3 years | 1.68 (0.94) | 1.38 (1.23)
Statistical Analysis 1: Comparison: Test Arm vs Control Arm; The concept of a "Visit" was developed by dividing the three-year-long observation interval into 3-month periods. All evaluations were mapped into 3-month-long bins (Reference: Mahapatra, S. et al. Autism Dev. Disord. 2018, 1). It was then hypothesized that there was a three-way interaction between an age group, Visit, and treatment. This hypothesis was modeled by applying the Linear Model with repeated measures, where a three-way interaction term was introduced to test the hypothesis; Test type: Other — Participants in the MITA group were matched to those in Control (treatment-as-usual) group using propensity score analysis based on age and all four ATEC subscales at baseline. Least squares means were calculated for all subscales at all visits; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 4.68

ADVERSE EVENTS:
Time Frame: Up to 3 years 6 months, on average 481 days
Arm/Group | Test Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/1009 | 0/1009
Serious Adverse Events (participants affected / at risk) | 0/1009 | 0/1009
Other Adverse Events (participants affected / at risk) | 0/1009 | 0/1009

LIMITATIONS AND CAVEATS:
The observational design of this study cannot definitively prove causality since unknown confounders may influence the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02708290/Prot_SAP_000.pdf